CLINICAL TRIAL: NCT06102343
Title: Open-label, Safety, and Efficacy Investigation on the Effects of ClearSkin Non-ablative ER: Glass 1540nm Laser Module in the Treatment of Acne Scars.
Brief Title: Safety and Efficacy Investigation on the Effects of ClearSkin Non-ablative ER:Glass 1540nm Laser Module in the Treatment of Acne Scars.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Alma Lasers (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALM-HAR-CLS-23-01
Record Dates: First submitted 2023-10-18; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Acne Scars - Mixed Atrophic and Hypertrophic
MeSH Terms: conditions — Hypertrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- acne scars treatment using the Alma Harmony platform with the ClearSkin applicator. (Experimental): treatment of acne scars using the ClearSkin non-ablative ER:Glass 1540nm laser Module.
  Interventions: Device: Alma Harmony

INTERVENTIONS:
Device: Alma Harmony — Acne scars treatment using non-ablative ER:Glass 1540 nm laser module.
  Other Names: ClearSkin applicator

SUMMARY:
The ClearSkin module, Er: Glass 1540nm, is largely used in the treatment of acne vulgaris and acne scars. The non-ablative ER:Glass 1540 nm laser deeply penetrates the skin, causing thermal damage to the sebaceous glands, destroying P. acnes bacteria and reducing sebum production, while leaving the epidermis intact. The integrated vacuum mechanism extracts accumulated sebaceous material from the pores, while contact cooling protects the skin, reducing pain and allowing for safer and more effective treatment of the sebaceous glands within the dermis. Based on this background, the investigators have considered a pilot study aimed at assessing the efficacy and safety of the ClearSkin Module in treating subjects with facial acne scars.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18 to 50 years
* Presence of mild to moderate facial acne scars (according to Goodman & Baron's scale)
* Subjects in reasonably good general health, according to the Investigator's judgment;
* Subjects who agree to avoid tanning during the entire investigational period;
* Subjects who agree to avoid any other facial procedure during the entire investigational period; including but not limited to: injectables or threads, peeling of any kind, dermabrasion, facial hair removal, or application of any cosmeceutical/pharmaceutical without the consent from the PI only.
* Subjects able to understand the full nature and the purpose of the investigation, including possible risks and side effects, able to cooperate with the Investigator and comply with the requirements of the entire investigation (ability to attend all the planned investigation visits according to the time limits included) based on Investigator's judgment.
* Subjects willing to sign an informed consent, consent to use their photos for future scientific or marketing purposes, according to the sponsor's needs.

Exclusion Criteria:

* Subjects with active infections
* Subjects with a history of keloid scarring or hypertrophic scar formation
* Subjects with previous medical treatment of the area, or oral retinoid drug prescribed within the past six months
* Subjects who have been tanning within the past 30 days;
* Previous surgical treatment of the area selected for the treatment with the investigational device;
* Subjects with any inflammatory skin condition e.g., eczema, active herpes simplex, etc. at the treatment site;
* Subjects with the presence of tattoos at the treatment site
* Subjects with skin cancer or any other cancer and/or any cancer drug therapy (such as ducabaxine, fluorouracil, methotrexate, etc.)
* Subjects with history of autoimmune disorder or evidence of immunosuppression;
* Subjects with collagen vascular diseases
* Subjects with thrombocytopenia
* Subjects with peripheral vascular disease
* Subjects with Melasma
* Pregnant or lactating subjects

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Reduction of at least 6 points in Goodman Baron's score at 3-month follow-up visit compared to baseline. | throughout the study, up to 1 year.
  comparison of acne scars' Goodman Baron's score at baseline with acne scars' Goodman Baron's score at 3-month follow-up visit compared to baseline.

SECONDARY OUTCOMES:
Improvement in the treated facial acne scars after ClearSkin according to the General Aesthetic Improvement Scale (GAIS), at the 3-month follow-up visit compared to baseline. | throughout the study, up to 1 year.
  70% of participants will demonstrate any improvement in the treated facial acne scars after ClearSkinTM according to the General Aesthetic Improvement Scale (GAIS), at the 3-month follow-up visit compared to baseline, as evaluated by three blinded assessors. The evaluation will be performed by means of the examination of the photography of treated facial acne scars performed using 2D photographs.
Improvement in the treated facial acne scars after ClearSkin according to the General Aesthetic Improvement Scale (GAIS), at the 1-month follow-up visit compared to baseline. | throughout the study, up to 1 year.
  Improvement in aesthetic appearance of the treated facial acne scars, as assessed by the principal investigator according to the General Aesthetic Improvement Scale (GAIS) at the 1-month follow-up visit compared to baseline. The evaluation will be performed by means of the examination of the photography of all treated facial acne scars performed using 2D photographs.
Improvement in skin texture of the treated facial acne scars. | throughout the study, up to 1 year.
  Improvement in skin texture of the treated facial acne scars, as evaluated by the 3D pictures taken at the 1- and 3-month follow-up visits compared to baseline.
Participant's satisfaction rates | throughout the study, up to 1 year.
  Participant's satisfaction with treatment with the investigational devices using a 5-point Likert scale, at 1- and 3-month follow-up visits.
Adverse Events frequency & intensity. | throughout the study, up to 1 year.
  Adverse Events frequency & intensity, occurring at any time during the trial or follow-up periods.
Pain level rates | throughout the study, up to 1 year.
  Pain level using NPRS, as evaluated at each treatment visit at the end of each treatment session.

CONTACTS AND LOCATIONS:
Overall Officials: Tiago Baptista, MD, Principal Investigator — Head of Up Clinic, Lisbon, Portugal
Locations (1):
- Up Clinic, Lisbon, Portugal